CLINICAL TRIAL: NCT06556732
Title: Potential Role of Eplerenone in Reducing Recurrence of Atrial Fibrillation in Patients With Structural Heart Disease
Brief Title: Role of Eplerenone in Reducing Recurrence of Atrial Fibrillation in Patients With Structural Heart Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelgaleel, Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Eplerenone in AF 2020
Record Dates: First submitted 2024-08-12; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study arm (Experimental): Were given Eplereone 25 mg daily
  Interventions: Drug: Eplereone
- Control arm (Placebo Comparator): Were given nothing
  Interventions: Drug: Eplereone

INTERVENTIONS:
Drug: Eplereone — Group A (study group): 50 patients received eplerenon 25 mg daily plus amiodarone and other medications not including non-dihydropyridine calcium channel blocker or digoxin.
  Other Names: Amiodarone

SUMMARY:
This is a prospective comparative study, conducted at Cardiology Department, Aswan University Hospital on AF patients with structural heart disease. Eplerenone 25 mg daily will be given and searching for AF recurrence among study population.

DETAILED DESCRIPTION:
This is a prospective comparative study, conducted at Cardiology Department, Aswan University Hospital, on 100 patients with AF and structural heart disease. AF is confirmed by electrocardiography. The patients were divided into 2 groups:

Group A (study group): 50 patients received eplerenon 25 mg daily plus amiodarone and other medications not including non-dihydropyridine calcium channel blocker or digoxin.

Group B (control group): 50 patients received amiodarone and other medications not including non-dihydropyridine calcium channel blocker or digoxin.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-valvular AF who underwent cardioversion to sinus rhythm either medical, electrical or even spontaneously

Exclusion Criteria:

* Patients with rheumatic heart disease.
* Thyroid dysfunction.
* Wolf-Parkinson-White (WPW) syndrome.
* Renal impairment.
* Hyperkalemia.
* Acute coronary syndrome.
* Pregnancy.
* Left ventricular (LV) dysfunction with ejection fraction (EF) less than 40%.
* On current use of eplerenone.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-10 (Estimated); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
AF recurrence | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Heart Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No